CLINICAL TRIAL: NCT02710214
Title: Effect of a Tissue Selective Estrogen Complex on Menopausal Symptoms in Women With MS: A Pilot Trial.
Brief Title: A TSEC for Symptom Management in Menopausal Women With Multiple Sclerosis
Acronym: MS-TSEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0512236
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Menopause; Multiple Sclerosis
Keywords: Hot flash; Estrogen; Women
MeSH Terms: conditions — Multiple Sclerosis; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duavee (Experimental): 1 Tablet of 0.45mg conjugated estrogens/20 mg bazedoxifene daily for 8 weeks
  Interventions: Drug: Tissue Selective Estrogen Complex
- Placebo (Placebo Comparator): Placebo pill daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tissue Selective Estrogen Complex — Once-daily dosing of Duavee for 8 weeks.
  Other Names: Duavee; TSEC
  Arms: Duavee
Drug: Placebo — Once-daily dosing of placebo for 8 weeks
  Arms: Placebo

SUMMARY:
Duavee is a hormone receptor modulator that has been approved for the treatment of menopausal symptoms in menopausal women. The goal of this 8-week randomized, double blind, placebo controlled pilot study, is to determine whether this medication alleviates menopausal symptoms in women with MS. The investigators will secondarily determine whether addressing menopausal symptoms ameliorates MS symptoms and, on MRIs, is not triggering worsening inflammation.

DETAILED DESCRIPTION:
Menopause in MS. Multiple sclerosis (MS) affects 3 times more women than men, and before age 50 in about 90% cases, i.e. prior to menopause. There is broad evidence for hormonal regulation of MS in animal models and in clinical cohorts. Around menopause, many clinical patients report symptom worsening associated with hot flashes, sleep disturbance or mood changes. Additionally, individuals at MS may be at increased risk of developing osteoporosis. Longer-term, an age-related decline in gonadal steroids might represent one sex-specific influence on the known age-related increases in disability and conversion to progressive course, which is marked by accelerated brain volume loss and neurodegeneration. Recent data suggest that MS disease severity may worsen after menopause.

* Hormone therapy (HT). Despite the benefits of HT (menopausal symptoms, bone density), very few women (<30% of our cohort) are currently taking HT for menopausal symptoms; this is a result of risks such as (1) breast and endometrial cancer, and (2) stroke in older women in the Women's Health Initiative. Recent data on HT use in MS (Nurses Health Study) did not show any adverse effects on MS course, and women who used HT reported better physical function than women who did not (Bove et al, Neurology 2016).
* Study Drug: Duavee, a tissue selective estrogen complex (TSEC), combines conjugated estrogens (CE) with the selective estrogen receptor modulator (SERM) bazedoxifene (BZA). BZA offsets estrogenic stimulation of endometrial and breast tissue, and CE 0.45mg/BZA 20mg is approved for menopausal symptom (hot flash) relief and osteoporosis prevention, with a favorable tolerability and safety profile.

In the current study, 24 women with MS and who are experiencing bothersome menopause symptoms will be enrolled and randomized to receive either 8 weeks of Duavee or 8 weeks of placebo. Visits will be: eligibility, baseline, and 2 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-62 years.
* Perimenopausal: 6 months of amenorrhea; women who had a bi-lateral oophorectomy; women without a uterus and who still have one or both ovaries, with FSH level > 20 mIU/mL and estradiol ≤ 50 pg/mL; women with a uterus who have skipped 2 or more menstrual cycles with an amenorrhea interval; women who are using the Mirena IUD or who have had an endometrial ablation and who still have one or both ovaries, with FSH level > 20 mIU/mL and estradiol ≤ 50 pg/mL
* Bothersome MS symptoms: Mean of two or more hot flashes/night sweats per 24 hrs; Hot flashes/night sweats rated as bothersome ('moderately' to 'a lot') and/or severe ('moderate' to 'severe') on 4 or more 12 hour (day/night) blocks of times
* In general good health (determined by medical history, blood pressure, and heart rate)
* No history of endometrial, ovarian, or breast cancer; No abnormal mammogram in the last 2 years; Absence of any current severe or unstable medical illness

MS considerations:

* If using psychotropic medications: no change in the past 3 months
* If on DMT, no change in past 6 months Normal vitamin D levels (20-50 ng/mL)

Exclusion Criteria:

* BMI >35 kg/m2 as higher BMI may affect PK/PD
* Use of hormone therapy or hormonal contraceptives 2 months prior to enrollment
* Use of any prescribed therapy that is taken specifically for hot flashes in the past 1 month.
* Use of any over-the-counter or herbal therapies that are taken specifically for hot flashes in the past 2 weeks.
* Use of selective estrogen receptor modulators (SERMs) or aromatase inhibitors during the 2 months before enrollment.
* Known hypersensitivity or contraindications to estrogen.
* Drug or alcohol abuse in the past 1 year
* Depression: moderate or severe (HAD score > 8) Other psychiatric disease meeting DSM-IV criteria
* Lifetime diagnosis of psychosis or bipolar disorder.
* Pregnancy, intending pregnancy, or breast feeding

History of any of the following, as determined by clinician review of the potential participant's medical history:

* Pre-breast cancer or high-risk breast cancer condition;
* Abnormal bleeding suggestive of endometrial pre-cancer;
* Endometrial hyperplasia;
* Asthma, diabetes mellitus, epilepsy, and migraine disorders that are not stable or under medical management;
* Active or past history of venous or arterial thromboembolism
* History of gallstones IF gallbladder intact
* Known or suspected estrogen-dependent neoplasia
* History of coronary artery disease
* Hypersensitivity (angioedema, anaphylaxis) to estrogens, bazedoxifene, or any ingredients
* Known hepatic impairment or disease
* Thyroid dysfunction on thyroid medications
* Known hypoparathyroidism
* Blood test results indicating:
* Liver function tests: AST >2.5 times upper limit of normal; ALT >2.5 times upper limit of normal; total bilirubin 1.5 times upper limit of normal;
* Kidney test: creatinine >1.5 mg/dL;
* Blood count: hematocrit <30%;
* Hemoglobin <8 g/dL.
* Current participation in another drug trial or intervention study.
* Inability or unwillingness to complete the study procedures.

MS considerations:

* Clinical relapse within the last three months (to ensure disease stability)
* Steroid treatment in prior 1 month
* Evidence of other structural brain disease (e.g. prior stroke)

MRI considerations:

* Metal implants
* Prior head trauma
* Claustrophobia requiring anxiolytic or sedation, or other contraindication to MRI.

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riley M Bove, MD, Principal Investigator — Assistant Professor of Clinical Neurology
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Bove R, Healy BC, Musallam A, Glanz BI, De Jager PL, Chitnis T. Exploration of changes in disability after menopause in a longitudinal multiple sclerosis cohort. Mult Scler. 2016 Jun;22(7):935-43. doi: 10.1177/1352458515606211. Epub 2015 Oct 7. PMID 26447063
- [Background] Bove R, Chitnis T, Houtchens M. Menopause in multiple sclerosis: therapeutic considerations. J Neurol. 2014 Jul;261(7):1257-68. doi: 10.1007/s00415-013-7131-8. Epub 2013 Oct 8. PMID 24101131
- [Background] Bove R, Healy BC, Secor E, Vaughan T, Katic B, Chitnis T, Wicks P, De Jager PL. Patients report worse MS symptoms after menopause: findings from an online cohort. Mult Scler Relat Disord. 2015 Jan;4(1):18-24. doi: 10.1016/j.msard.2014.11.009. Epub 2014 Dec 9. PMID 25787049
- [Background] Bebo BF Jr, Dehghani B, Foster S, Kurniawan A, Lopez FJ, Sherman LS. Treatment with selective estrogen receptor modulators regulates myelin specific T-cells and suppresses experimental autoimmune encephalomyelitis. Glia. 2009 May;57(7):777-90. doi: 10.1002/glia.20805. PMID 19031437
- [Background] Boccardi M, Ghidoni R, Govoni S, Testa C, Benussi L, Bonetti M, Binetti G, Frisoni GB. Effects of hormone therapy on brain morphology of healthy postmenopausal women: a Voxel-based morphometry study. Menopause. 2006 Jul-Aug;13(4):584-91. doi: 10.1097/01.gme.0000196811.88505.10. PMID 16837880
- [Background] Bove R, Secor E, Chibnik LB, Barnes LL, Schneider JA, Bennett DA, De Jager PL. Age at surgical menopause influences cognitive decline and Alzheimer pathology in older women. Neurology. 2014 Jan 21;82(3):222-9. doi: 10.1212/WNL.0000000000000033. Epub 2013 Dec 11. PMID 24336141
- [Background] North American Menopause Society. The 2012 hormone therapy position statement of: The North American Menopause Society. Menopause. 2012 Mar;19(3):257-71. doi: 10.1097/gme.0b013e31824b970a. PMID 22367731
- [Background] Pozzilli C, De Giglio L, Barletta VT, Marinelli F, Angelis FD, Gallo V, Pagano VA, Marini S, Piattella MC, Tomassini V, Pantano P. Oral contraceptives combined with interferon beta in multiple sclerosis. Neurol Neuroimmunol Neuroinflamm. 2015 Jun 18;2(4):e120. doi: 10.1212/NXI.0000000000000120. eCollection 2015 Aug. PMID 26140279
- [Background] Voskuhl RR, Wang H, Wu TC, Sicotte NL, Nakamura K, Kurth F, Itoh N, Bardens J, Bernard JT, Corboy JR, Cross AH, Dhib-Jalbut S, Ford CC, Frohman EM, Giesser B, Jacobs D, Kasper LH, Lynch S, Parry G, Racke MK, Reder AT, Rose J, Wingerchuk DM, MacKenzie-Graham AJ, Arnold DL, Tseng CH, Elashoff R. Estriol combined with glatiramer acetate for women with relapsing-remitting multiple sclerosis: a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Jan;15(1):35-46. doi: 10.1016/S1474-4422(15)00322-1. Epub 2015 Nov 29. PMID 26621682
- [Derived] Morales-Rodriguez D, Anderson A, Nylander A, Hsu S, Singh J, Rowles W, Walsh CM, Braley TJ, Bove R. Well-being at midlife: Correlates of mental health in ambulatory menopausal women with multiple sclerosis. Mult Scler. 2023 Oct;29(11-12):1493-1502. doi: 10.1177/13524585231197056. Epub 2023 Sep 16. PMID 37715710

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duavee | Placebo
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duavee | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (4.2) | 50.8 (2.9) | 51.2 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Disease Modifying Therapy (DMT) [Count of Participants; unit: Participants]
  None | 1 | 5 | 6
  Glatiramer Acetate | 1 | 2 | 3
  Interferons | 1 | 0 | 1
  Teriflunomide | 1 | 0 | 1
  Fingolimod | 3 | 2 | 5
  Dimethyl Fumarate | 1 | 1 | 2
  Ocrelizumab | 3 | 1 | 4
  Rituximab | 0 | 1 | 1
  Natalizumab | 1 | 0 | 1
Expanded Disability Status Scale Score [Median (Inter-Quartile Range); unit: units on a scale] — Scale of 0 to 10 (higher scores indicate greater disability).
  units on a scale | 3.0 [2.5 to 4.0] | 3.0 [2.0 to 6.0] | 3.0 [2.5 to 4.5]
Timed 25 Foot Walk [Mean (Standard Deviation); unit: seconds] — Population: N=16 with available data.
  seconds
    number analyzed (Participants) | 7 | 9 | 16
    (all) | 4.91 (0.7) | 5.33 (1.6) | 5.15 (1.3)
Symbol Digit Modalities (SDMT) Raw Score [Median (Inter-Quartile Range); unit: number of correct responses] — The Symbol Digit Modalities Test (SDMT) is a screening instrument commonly used in clinical and research settings to assess cognitive dysfunction in MS. The final score is the correct number responses completed in 90 seconds and scores range between 0 and 110; higher scores indicate better performance.
  number of correct responses | 43.5 [33 to 53] | 44 [37 to 52] | 44 [37 to 52]
SDMT (z-score) [Median (Inter-Quartile Range); unit: z-score] — Regression-based norms for the SDMT were used to convert participants' raw scores to demographically adjusted Z-scores, correcting for the effects of age, gender, and education. Scores are normalized so that 0 represents the mean, scores above 0 fall above the mean and are associated with greater performance on the SDMT. Scores below 0 fall below the mean and are associated with poorer performance on the SDMT
  z-score | -0.91 [-1.65 to 0.19] | -0.93 [-1.76 to 0.07] | -0.92 [-1.66 to 0.07]
Letter Number Sequencing (LNS) [Median (Inter-Quartile Range); unit: number of correct responses] — The Letter Number Sequencing (LNS) is administered to asses working memory and processing speed. The score range is 0 to 21; higher scores indicate better performance on this test.
  number of correct responses | 10.5 [10 to 12] | 9.5 [8.5 to 11] | 10 [9 to 11]
Multiple Sclerosis Quality of Life 54 (MSQOL-54) [Median (Inter-Quartile Range); unit: units on a scale] — Score range 0 to 100 for each sub-scale (mental, physical, energy); higher scores indicate better quality of life within that domain. Population: N=20 with available data.
  units on a scale
    MSQOL-54 Mental: number analyzed (Participants) | 11 | 9 | 20
    MSQOL-54 Mental | 79.3 [72.6 to 82.3] | 71.5 [49 to 86] | 74.2 [67.5 to 85.1]
    MSQOL-54 Physical: number analyzed (Participants) | 11 | 9 | 20
    MSQOL-54 Physical | 64.3 [51.4 to 78.0] | 45.8 [39.1 to 76.7] | 63.0 [44.4 to 76.8]
    MSQOL-54 Energy: number analyzed (Participants) | 11 | 9 | 20
    MSQOL-54 Energy | 36 [24 to 76] | 40 [12 to 52] | 38 [20 to 60]
Multiple Sclerosis Rating Scale Composite Score [Median (Inter-Quartile Range); unit: units on a scale] — Score range of 0 to 32 (higher scores indicate worse patient reported disability). Population: N=20 with available data.
  units on a scale
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 6 [3 to 10] | 11 [5 to 16.5] | 8.5 [3 to 12.5]
Multiple Sclerosis Neuropsychological Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Score range 0 to 60 (scores >27 indicate cognitive impairment). Population: N=20 with available data.
  units on a scale
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 16 [5 to 35] | 27 [18 to 35] | 19.5 [11.5 to 34]
Bladder Control Score [Median (Inter-Quartile Range); unit: units on a scale] — Score range of 0 to 12 (higher scores indicate greater bladder dysfunction). Population: N=20 with available data.
  units on a scale
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 1 [0 to 5] | 2 [0 to 7] | 1.5 [0 to 4.5]
Hot Flashes (per 24 hours) [Median (Inter-Quartile Range); unit: hot flashes/day] — Median calculated from 2 weeks of daily hot flash diaries. Population: N=19 with available data.
  hot flashes/day
    number analyzed (Participants) | 9 | 10 | 19
    (all) | 5.6 [2.2 to 8.9] | 3.4 [1.6 to 8.6] | 4.1 [1.8 to 8.6]
Hot Flash Related Daily Interference Scale [Median (Inter-Quartile Range); unit: units on a scale] — Score range 0 to 100 (higher scores indicate greater interference of hot flashes with daily life). Population: N=16 with available data.
  units on a scale
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 22 [7 to 26.5] | 27 [15.5 to 66.5] | 23.5 [9.5 to 31.7]
Insomnia Severity Index [Median (Inter-Quartile Range); unit: units on a scale] — Score range of 0 to 28 (0-7 indicates no clinically significant insomnia, 8-14 indicates sub-threshold insomnia, 15-21 indicates clinical insomnia of moderate severity, and 22-28 indicates severe clinical insomnia). Population: N=9 with available data.
  units on a scale
    number analyzed (Participants) | 4 | 5 | 9
    (all) | 10.5 [8.2 to 16.5] | 8 [7.5 to 21] | 9 [8 to 16.5]

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Related Daily Interference Scale (HFRDIS) Score
Description: The interference of vasomotor symptoms (VMS) with daily life will be assessed using the HFRDIS. Scores range from 0 to 100; higher scores indicate greater interference of hot flashes with daily life.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 21 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | 4 [0.5 to 14] | 9 [0 to 33]

2. Primary Outcome: Change in Number of Participants Who Experienced a Reduction in Hot Flashes Per 24 Hours From Baseline to 8 Weeks
Description: The number of daily vasomotor symptoms (VMS) will be collected in the form of hot flashes per 24 hours. The average hot flashes per day will be determined at 2 week intervals (baseline, 2 weeks, 4 weeks, and 8 weeks). The number of women experiencing reduction in hot flashes at week 8 compared to baseline will be counted; when baseline data is unavailable 1-2 week on study data will be used.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 18 participants, due to missing data; in 3 cases, weeks 1-2 of on- study data was used when baseline was unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 9
Participants | 9 | 8

3. Primary Outcome: Change in Average Hot Flashes Per Day From Baseline to 8 Weeks
Description: The number of daily vasomotor symptoms (VMS) will be collected in the form of hot flashes per 24 hours. The average hot flashes per day will be determined at 2 week intervals (baseline, 2 weeks, 4 weeks, and 8 weeks). The average reduction in hot flashes per day over the course of the trial will be determined from the difference between 8 week and baseline frequency (by randomization group, treatment or placebo). When baseline data is not available, the 2 weeks on study data will be used as 'baseline'. Differences <0 indicate reduction in hot flash frequency over the course of the trial.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 21 participants, due to missing data; in 3 cases, weeks 1-2 of on- study data was used when baseline was unavailable.
Measure: Median (Inter-Quartile Range); unit: hot flashes/day
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 10 | 11
hot flashes/day | -2.1 [-3.8 to 0.3] | -2.6 [-7.1 to -0.6]

4. Primary Outcome: Number of Participants Reporting Side Effects on the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The primary measure will be the percentage of subjects reporting side effects (yes or no) on the Satisfaction Questionnaire for Medication (TSQM). The TSQM is used to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction.
Time Frame: 8 weeks
Population: Data for this measure available only for 16 participants, due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 2 | 1

5. Primary Outcome: Change in the Expanded Disability Status Scale (EDSS)
Description: EDSS total score is a metric used for quantifying disability in MS and monitoring changes in the level of disability over time. The EDSS will be assessed by a the trial neurologist at baseline and end of study (8 weeks). The score range is 0 to 10; higher scores indicate greater disability. All analyses were performed according to the intention-to-treat principle (primary) then the per-protocol principle.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 22 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | -0.5 [-0.5 to 0] | 0 [-0.5 to 0]

6. Secondary Outcome: Change in the MS Quality of Life 54 (MSQOL-54)
Description: MS Quality of Life 54 (MSQOL-54) composite scores provide a patient reported quality of life score assessing physical QOL and mental QOL. A sub-scale of this assessment also assesses energy QOL. These will be measured at baseline and end of study (8 weeks). These scores fall within the range of 0 to 100; higher scores indicate better QOL within that domain or sub-scale.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 16 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 7
units on a scale
  MSQOL-54: Physical | 5.2 [-2.2 to 9.8] | 0 [-3.2 to 17.8]
  MSQOL-54: Mental | 0.3 [-2.8 to 3.8] | 0 [-14.1 to 11.7]
  MSQOL-54: Energy | 0 [-6 to 6.5] | 0 [-12 to 32]

7. Secondary Outcome: Change in the Bladder Control Scale (BLCS)
Description: Bladder function will be assessed using the BLCS. Patient reported scores will be collected at baseline and at the end of study (8 weeks); scores fall within the range of 0 to 12. Higher scores indicate worse bladder function.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 16 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 7
units on a scale | 1 [0 to 2.5] | 0 [0 to 2.5]

8. Secondary Outcome: Change in the Multiple Sclerosis Rating Scale (MSRS)
Description: Patient reported disability will be measured by the MSRS at baseline and end of study (8 weeks). Scores range of 0 to 32; higher scores indicate worse patient reported disability.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 16 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 7
units on a scale | 1 [-2.5 to 1.5] | 0 [-1 to 2]

9. Secondary Outcome: Change in the Multiple Sclerosis Neuropsychological Questionnaire (MSNQ)
Description: Cognitive function will be assessed by the MSNQ at baseline and end of study (8 weeks). Scores range 0 to 60 (scores >27 indicate cognitive impairment).
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 16 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 9 | 7
units on a scale | -2 [-4 to 0] | 0 [-4 to 0]

10. Secondary Outcome: Change in the Symbol Digit Modalities Test (SDMT) Raw Score
Description: SDMT is a screening instrument commonly used in clinical and research settings to assess cognitive dysfunction in MS. The SDMT will be administered at baseline and end of study (8 weeks). The final raw score is the correct number responses completed in 90 seconds and scores range between 0 and 110; higher scores indicate better performance.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 21 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale | 3 [2 to 10] | 1 [-3 to 2.25]

11. Secondary Outcome: Change in SDMT Z-score
Description: Regression-based norms for the SDMT were used to convert participants' raw scores at baseline and end of study (8 weeks) to demographically adjusted Z-scores, correcting for the effects of age, gender, and education. Scores are normalized so that 0 represents the mean, scores above 0 fall above the mean and are associated with greater performance on the SDMT. Scores below 0 fall below the mean and are associated with poorer performance on the SDMT.
Time Frame: Baseline and 8 weeks
Population: N=21 with available data.
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 11 | 10
z-score | 0.39 [-0.18 to 1.01] | 0.13 [-0.30 to 0.26]

12. Secondary Outcome: Change in Letter Number Sequencing (LNS) Performance
Description: The LNS is administered to asses working memory and processing speed at baseline and end of study (8 weeks). The score range is 0 to 21; higher scores indicate better performance on this test.
Time Frame: Baseline and 8 weeks
Population: Data for this measure available only for 21 participants, due to missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale | 0 [0 to 1] | 1 [0 to 2]

13. Secondary Outcome: Number of Participants With New or Enhancing Lesions on MRI
Description: To verify that CE+BZA does not yield any marked changes in inflammatory activity, a randomized subset of 12 participants will undergo MRI at baseline and end of study (8 weeks) to evaluate for new T2 lesions and new gadolinium enhancing lesions.
Time Frame: 8 weeks
Population: N=12 with MRI; participants were randomized to the MRI or no MRI group in this double blinded study; thus, by chance a higher number of women allocated to the Duavee arm received MRI's.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 8 | 4
Participants | 0 | 1

14. Secondary Outcome: Number of Missed Doses
Description: The number of missed doses will be assed at the end of study visit.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: missed doses
Arm/Group | Duavee | Placebo
Number analyzed (Participants) | 11 | 10
missed doses | 0 [0 to 0] | 1 [0 to 9]

ADVERSE EVENTS:
Time Frame: 8 weeks, from start of study medication (at baseline visit) to end of study visit.
Arm/Group | Duavee | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Planned low sample size and our pre-specified power calculation allowed 80% power to observe a greater mean change in the treatment than in the control arm but did not provide sufficient power to assess statistical significance in this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT02710214/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02710214/SAP_001.pdf